CLINICAL TRIAL: NCT01588392
Title: Effects of Short Bouts of Physical Activity in Low-income Preschool-age Children
Brief Title: Short bouTs of Exercise for Preschool-age Children
Acronym: STEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Amherst (Other)
Responsible Party: Principal Investigator, Sofiya Alhassan, Assistant Professor, University of Massachusetts, Amherst
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2010-0817
Record Dates: First submitted 2012-04-25; First posted 2012-05-01 (Estimated); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Physical Activity
Keywords: Physical activity; preschoolers
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Short bouts of structured activity (Experimental)
  Interventions: Behavioral: Short bouts of structured physical activity
- Unstructured physical activity (Active Comparator)
  Interventions: Behavioral: Unstructured physical activity

INTERVENTIONS:
Behavioral: Short bouts of structured physical activity — Short bouts of structured physical activity preschools will be asked to implement age-appropriate 10 minute structured physical activity routines within the classroom setting followed by 20 minutes of usual unstructured playtime activities. Intervention will be implemented for a total of 30 minutes during both morning and afternoon gross motor playtime 5 days/week for 6 months.
  Other Names: Instant Recess for preschoolers
  Arms: Short bouts of structured activity
Behavioral: Unstructured physical activity — Unstructured physical activity intervention will consist of 30 minutes of supervised unstructured free playtime twice. intervention will be delivered during both morning and afternoon gross motor playtime for 5 days/week for 6 months.
  Other Names: Free playtime
  Arms: Unstructured physical activity

SUMMARY:
The purpose of this study is to examine if short bouts of structured physical activity implemented within the classroom setting as part of designated gross-motor playtime will increase preschool-age children during-school physical activity level.

DETAILED DESCRIPTION:
Most preschool centers provide two 30-minute sessions of gross-motor/outdoor playtime per preschool day. Within this time frame, children accumulate most of their activity within the first 10 minutes. This study is a cluster randomized controlled study designed to examine the effects of short bouts of structured physical activity implemented within the classroom setting as part of designated gross-motor playtime on during-school physical activity in preschoolers. Results from this intervention could provide evidence that a physical activity policy that exposes preschoolers to shorter bouts of structured physical activity throughout the preschool day could potentially increase preschooler's physical activity levels.

ELIGIBILITY:
Inclusion Criteria:

* Attend one of 10 participating preschool centers
* Attend preschool full-time
* Children between 2.9 - 5 years of age on the date of baseline assessment

Exclusion Criteria:

* Did not have a condition limiting their participation in routine gross-motor playtime at preschool
* Unable to wear the activity monitor

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 323 (Actual)
Dates: Start 2011-11; Primary Completion 2013-05 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Physical activity levels at 6-month | Baseline, 3-month and 6-month after study initiation
  Physical activity levels will be assessed with accelerometer and direct observation system

CONTACTS AND LOCATIONS:
Overall Officials: Sofiya Alhassan, Principal Investigator — University of Massachusetts, Amherst
Locations (1):
- Preschool centers in Springfield, MA, Springfield, Massachusetts, United States

REFERENCES:
- [Derived] Alhassan S, Nwaokelemeh O, Mendoza A, Shitole S, Whitt-Glover MC, Yancey AK. Design and baseline characteristics of the Short bouTs of Exercise for Preschoolers (STEP) study. BMC Public Health. 2012 Aug 1;12:582. doi: 10.1186/1471-2458-12-582. PMID 22853642